CLINICAL TRIAL: NCT04096950
Title: A Study to Investigate the Safety, Tolerability , Pharmacokinetics of Single Ascending Dose of MT-3921 in Subjects With Acute Spinal Cord Injury
Brief Title: Safety and Pharmacokinetics Study of MT-3921 in Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-3921-G01
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MT-3921 (Experimental): Intravenous, single dose
  Interventions: Biological: MT-3921 Low dose

INTERVENTIONS:
Biological: MT-3921 Low dose — MT-3921 Low dose, intravenous, single dosing

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of MT-3921 in subjects with spinal cord injury.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single ascending dose study of MT-3921 in subjects with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

Additional screening criteria check may apply for qualification:

* Provide written informed consent prior to beginning any study procedures
* Cervical spinal cord injury, ASIA impairment scale grade A, B, and C with the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Neurological level of injury between C4 and C8
* Male or female subjects aged between 18 and 65 years
* Body mass index (BMI) <35
* Has had stabilization surgery (if needed) following their SCI and prior to receiving MT-3921

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

* Any concomitant injury that interferes with the performance, interpretation or validity of neurological examinations
* Poly-traumatic Injury as defined by Injury Severity Score (ISS) values > 25
* Penetrating spinal cord injuries
* Traumatic transection of the spinal cord or spinal cord contusion size > 3 cm determined by MRI
* Any other significant pre-existing medical conditions prior to spinal cord injury or current conditions that, in the judgement of the iInvestigator, may increase the risks associated with study participation
* Subjects with HIV, HBV or HCV positive
* Psychoactive substance use disorder
* History or presence of malignancy within the last 5 years prior to screening
* Pregnant or nursing women
* Subjects with hereditary fructose intolerance
* History of anaphylaxis or significant allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-04-19 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with adverse events within 6 months after single injection of MT-3921 | 6 Months

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile (Cmax) | 6 months post-dose
  PK samples will be collected at 0, 1, 4, 8 hours, 1, 2, 7 days, and 1, 2, 3, 6 months post-dose.
PK profile (tmax) | 6 months post-dose
  PK samples will be collected at 0, 1, 4, 8 hours, 1, 2, 7 days, and 1, 2, 3, 6 months post-dose.
PK profile (t½) | 6 months post-dose
  PK samples will be collected at 0, 1, 4, 8 hours, 1, 2, 7 days, and 1, 2, 3, 6 months post-dose.
PK profile (AUC) | 6 months post-dose
  PK samples will be collected at 0, 1, 4, 8 hours, 1, 2, 7 days, and 1, 2, 3, 6 months post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Development,, Study Director — Tanabe Pharma America, Inc.
Locations (13):
- United States (13):
  - UC Davis Medical Center, Sacramento, California
  - Northwestern University / Shirley Ryan Ability LAB (SRALAB), Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Carolinas Healthcare System / Atrium Health, Charlotte, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - VA Commonwealth Univ. School of Medicine, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided